CLINICAL TRIAL: NCT05494593
Title: An Open-label, Multicenter, Phase 4 Study to Assess the Effects of a Prophylactic Immune Tolerizing Regimen in MPS II Treatment-Naïve Patients Planned to Receive ELAPRASE Who Are at Risk of Developing Persistent Neutralizing Antibodies
Brief Title: A Study of ELAPRASE in Treatment-naïve Participants With Hunter Syndrome (Mucopolysaccharidosis [MPS] II)
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was closed due to enrollment challenges
Sponsor: Takeda (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-665-4003
Record Dates: First submitted 2022-08-08; First posted 2022-08-10 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Mucopolysaccharidosis (MPS); Hunter Syndrome
MeSH Terms: conditions — Mucopolysaccharidoses; Mucopolysaccharidosis II | interventions — idursulfase; Rituximab; Methotrexate; Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- ITR + ELAPRASE (Experimental): Participants will receive prophylactic ITR which consist of rituximab, methotrexate and IVIG in a 5-week cycle. Following the completion of 1 cycle and at the Month 6, 12, and 18 study visits, an assessment will be made regarding the need for administering another 5-week cycle of the ITR depending on the trend of the participants anti-idursulfase antibody titers and lymphocyte quantitation and CD19 percent (%) recovery.
  Elaprase treatment (IV, weekly) will start 1 day after the initiation of the first cycle of ITR and continue for 104 weeks.
  The dose of ELAPRASE will be calculated based on the participant's weight at each visit.
  Interventions: Drug: ELAPRASE; Drug: Rituximab; Drug: Methotrexate; Drug: Intravenous Immunoglobulin (IVIG)

INTERVENTIONS:
Drug: ELAPRASE — Participants will receive 0.5 milligram per kilogram (mg/kg) of body weight of ELAPRASE, intravenous, infusion for 104 weeks.
  Other Names: Idursulfase
Drug: Rituximab — Participants will receive 375 milligram per square meter per dose (mg/m^2/dose) of intravenous rituximab weekly for 4 weeks in 5-week cycle.
Drug: Methotrexate — Participants will receive 0.4 mg/kg of methotrexate by mouth (PO) 3 times per week for 5 weeks in each cycle.
Drug: Intravenous Immunoglobulin (IVIG) — Participants will receive 500 mg/kg of IVIG every 4 weeks in 5-week cycle.

SUMMARY:
The main aim of this study is to evaluate the ability of a prophylactic immune tolerizing regimen (ITR) to prevent or reduce the development of high titer anti-idursulfase antibodies in treatment-naïve participants with Hunter syndrome.

In this open label, single arm study, all participants will receive ELAPRASE treatment and a prophylactic ITR.

Participants will be treated with ELAPRASE for up to 104 weeks. The prophylactic ITR will start 1 day prior to the start of ELAPRASE. The prophylactic ITR will consist of a 5-week cycle of: Rituximab (intravenously [IV], weekly for 4 weeks); Methotrexate (oral, 3 times per week for 5 weeks) and intravenous immunoglobulin (IVIG) (IV, every 4 weeks of the cycle).

Following the completion of 1 cycle, an assessment will be made at Month 6, 12, and 18 regarding the need for administering another 5-week cycle of the ITR.

Participants will be in the study for approximately 112 weeks (including 6 weeks for screening, up to 104 weeks for treatment, and 2 weeks for follow-up).

ELIGIBILITY:
Inclusion Criteria:

* Participant is male.
* Participant is ELAPRASE-naïve at study entry.
* Participant must have a documented diagnosis of MPS II. The following combination will be accepted as diagnostic of MPS II:

  * Participant has a deficiency in iduronate-2-sulfatase (I2S) enzyme activity of less than or equal to (<=) 10 percent (%) of the lower limit of the normal range as measured in plasma, fibroblasts, or leukocytes (based on the reference laboratory's normal range). The participant has a normal enzyme activity level of at least 1 other sulfatase as measured in plasma, fibroblasts, or leukocytes (based on the reference laboratory's normal range).
  * Participant has a documented mutation in the IDS gene; additionally, participants must have a severe mutation (example, large deletion or complex gene rearrangement), which is predicted to lead to development of a persistent anti-idursulfase antibody response.
* Participant will be less than (<) 6 years of age at enrollment.
* Participant has a negative test result for serum anti-idursulfase antibodies.

Exclusion Criteria:

* Participant has received treatment with any investigational drug within the 30 days prior to study entry.
* Participant has received or is receiving treatment with idursulfase-IT.
* Participant has received growth hormones, a cord blood infusion, or a bone marrow transplant at any time.
* Participant has received blood product transfusions within 90 days prior to screening.
* Participant is unable to comply with the protocol as determined by the investigator.
* Participant has known or suspected intolerance or hypersensitivity to the investigational product(s), closely related compounds, or any of the stated ingredients, including the prophylactic ITR.
* Participant has current or recurrent disease that could affect the action, absorption, or disposition of the investigational product, or clinical or laboratory assessments.
* Participant has current or relevant history of physical or psychiatric illness, or any medical disorder that may require treatment or make the participant unlikely to fully complete the study, or any condition that presents undue risk from the investigational product or procedures.
* Participant has current use of any medication (including over-the-counter, herbal, or homeopathic preparations) that could affect (improve or worsen) the condition being studied, or could affect the action, absorption, or disposition of the investigational product(s), or clinical or laboratory assessment (Current use is defined as use within 30 days).
* Within 30 days prior to the first dose of investigational product, the participant has been enrolled in a clinical study (including vaccine studies) that, in the investigator's opinion, may impact this study.

Max Age: 6 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2025-08-29 (Actual); Study Completion 2025-08-29 (Actual)

PRIMARY OUTCOMES:
Rate of Anti-Idursulfase Antibodies Formation, Including Anti-Idursulfase Antibodies That Have Enzyme Neutralizing Activity | Up to 24 months
  Serum samples will be collected for evaluation of anti-idursulfase antibodies including binding antibodies and neutralizing antibodies. Analysis of anti-idursulfase antibodies will be conducted using validated 3-tier immunoassay methods. Rate will be defined as the number of participants having positive antibodies compared to the total number of participants.

SECONDARY OUTCOMES:
Correlation Between Anti-drug Antibody (ADA) Responses and Iduronate-2-Sulfatase (IDS) Gene Mutations and Clinical Outcomes | Every 6 months up to 24 months
  Correlation between ADA responses and IDS gene mutations and clinical outcomes (efficacy and safety) every 6 months in comparison to historical results from Study SHPELA- 401 (NCT02455622) without immune tolerance treatment will be reported. Analysis of covariance will be performed to correlate ADA response, IDS gene mutation and clinical outcomes.
Change From Baseline in Urinary Glycosaminoglycan (uGAG) Levels Normalized to Urine Creatinine | Up to 24 months
  Urine samples will be collected for the determination of uGAG levels and urine creatinine monthly prior to dosing. Change from baseline in uGAG levels normalized to urine creatinine will be reported.
Change From Baseline in Normalized uGAG per Upper Limit of Normal for age (uGAG)/ULN) | Up to 24 months
  Urine samples will be collected for the determination of uGAG levels monthly prior to dosing. Change from baseline in normalized uGAG/ULN will be reported.
Change From Baseline in Liver Volume | Up to 24 months
  Liver volume will be measured using abdominal ultrasonography. Change from baseline values for liver volume will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (8):
- United States (8):
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Rady Childrens Hospital San Diego - PIN, San Diego, California
  - The Lundquist Institute for BioMedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Ann and Robert H Lurie Childrens Hospital of Chicago, Chicago, Illinois
  - Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - NewYork-Presbyterian Morgan Stanley Children's Hospital, New York, New York
  - The Cleveland Clinic Foundation, Twinsburg, Ohio

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as there is a reasonable likelihood that individual participants could be re-identified (due to the limited number of study participants)

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/15c973b2efde4ff6?idFilter=%5B%22TAK-665-4003%22%5D